CLINICAL TRIAL: NCT03944564
Title: Kognitivne in Gibalne Prednosti stoječega Delovnega Mesta (KOGIS)
Brief Title: Cognitive and Motor Benefits of Standing
Acronym: KOGIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Science and Research Centre Koper (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KOGIS
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Pain, Acute; Muscle Tone Abnormalities; Work-Related Condition; Sensory Deficit
Keywords: cognition; brain activity; cognitive reserve; work productivity; musculoskeletal discomfort; attention
MeSH Terms: conditions — Acute Pain | interventions — Sitting Position

STUDY DESIGN:
Intervention Model Description: Randomized, controlled crossover trial
Masking Description: Participants will receive a general information about the study protocol and received three conditions in a random order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition 1: sitting (Active Comparator): Four hours of sitting condition will be applied with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales will be monitored.
  Interventions: Behavioral: Sitting
- Condition 2: static standing (Active Comparator): Four hours of static standing condition will be applied with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales will be monitored.
  Interventions: Behavioral: Static standing
- Condition 3: dynamic standing (Active Comparator): Four hours of static standing condition will be applied with ad-libitum breaks for toilet use and stretching. During this condition all cognitive, motor and pain scales will be monitored.
  Interventions: Behavioral: Dynamic standing

INTERVENTIONS:
Behavioral: Sitting — We propose a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions will be applied: 4 hours of sitting, static standing and dynamic standing. Both standing conditions will be done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: SIT
  Arms: Condition 1: sitting
Behavioral: Static standing — We propose a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions will be applied: 4 hours of sitting, static standing and dynamic standing. Both standing conditions will be done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: STAT
  Arms: Condition 2: static standing
Behavioral: Dynamic standing — We propose a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification. To evaluate this form on healthy subjects, three different conditions will be applied: 4 hours of sitting, static standing and dynamic standing. Both standing conditions will be done with height-adjustable table which was developed at the University of Michigan (Ann Arbor, Michigan, USA)
  Other Names: DYN
  Arms: Condition 3: dynamic standing

SUMMARY:
Upright-working has been proven to benefit health by combating the negative effects of physical inactivity. However, long-term commitment to static standing regimens may be limited due to symptoms of musculoskeletal fatigue that may develop during prolonged static standing in the absence of facilitated weight shifting. We propose a dynamic standing approach (working while standing accompanied by small periodic stepping movements) as a more tolerable and thereby more applicative lifestyle modification.

DETAILED DESCRIPTION:
Within-group design to study the effects of standing-and-working accompanied by periodic movement compared to standing-and-working and to sitting-and-working on measures of musculoskeletal fatigue and discomfort, and physiological measures, in healthy normal control subjects, middle-aged to older adults. Measures of musculoskeletal and subjective discomfort and fatigue will be assessed in three sessions, i.e. "seated", "static standing", and "dynamic standing" (see below). During these test sessions subjects will perform small assignments using a computer mimicking light office work, including several tests measuring attention span. The first session will be the seated condition for all participants. Sessions 2 and 3 will be randomized between static or dynamic standing.

Prior to any research procedures, written informed consent will be obtained from each subject followed by initial study eligibility screening. Eligibility screening includes clinical screening questions, including, but not limited to, questions regarding significant history of cardiovascular disease, history of lower extremity pain and fractures, back pain, and migraines.

Subjects will stand behind a height adjustable table that is positioned about 0.5 meters from a wall. For the "static standing" position subjects will be asked to stand behind the table. No specific restrictions for standing will be imposed on subjects (e.g. "do not move" or "stand quietly"). For the "dynamic standing" condition participants will stand behind the same table but received periodic cues to induce weight-shifting steps. A seated control session condition will also be used to get baseline musculoskeletal subjective ratings for the same time period. Each sitting or standing session will not exceed 4 hour. As many rest breaks will be provided to the subject as needed. The entire test session may take up to approximately 5 hours.

The experimental testing protocol will be conducted preferably in the morning over three or more different days. Each day will be dedicated to one testing condition. Subjects will stand on an anti-fatigue mat during the static and dynamic standing sessions. For the standing conditions, rest breaks (e.g. sitting or walking around) will be provided as needed. During the study session caffeine consumption will be prohibited in order to standardize the stimulant effect of caffeine across subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (both gender, age range 18-64 years) who are currently employed.

Exclusion Criteria:

1. Inability to stand or walk without an assistive device
2. History of symptoms in stance that preclude safe and comfortable participation, such as dizziness and lightheadedness, orthostasis, severe symptomatic leg or back musculoskeletal pain, or medication side effects
3. History of symptomatic cardiovascular or pulmonary disease
4. History of rheumatic arthritis
5. History of stroke or other neurologic conditions with residual sensorimotor deficits
6. History of chronic pain syndrome requiring narcotic analgesics
7. Neurological disorders
8. Evidence of dementia
9. Diabetics: low or poorly controlled blood glucose
10. Any other history of medical or psychiatric comorbidity precluding safe participation in the project

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall movement - accelerometry | change in activity levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Overall movement (counts/min)
Musculoskeletal discomfort | change in musculoskeletal discomfort levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Rate of total musculoskeletal discomfort development (mm/min)
Leg swelling | change in leg swelling levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Average swelling for both legs (cm)

SECONDARY OUTCOMES:
Oxygen uptake | change in oxygen consumption between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Oxygen uptake VO2 (ml/min/kg)
Attention levels | change in attentional levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Measuring attention with Stroop test (seconds)
Executive control | change in executive control and cognitive switching levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  Executive functions measured with TMT test (seconds)
Brain electrocortical activity | change in electrocortical activity levels between all three conditions, which will be measured on average 3 days in-between (maximum length of measurements per subject = 15 days)
  EEG measurements (frequency analysis and ERP analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Science and research centre Koper, Koper, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Background] Levine JA, Schleusner SJ, Jensen MD. Energy expenditure of nonexercise activity. Am J Clin Nutr. 2000 Dec;72(6):1451-4. doi: 10.1093/ajcn/72.6.1451. PMID 11101470
- [Background] Levine JA, Kotz CM. NEAT--non-exercise activity thermogenesis--egocentric & geocentric environmental factors vs. biological regulation. Acta Physiol Scand. 2005 Aug;184(4):309-18. doi: 10.1111/j.1365-201X.2005.01467.x. PMID 16026422
- [Background] Hamilton MT, Hamilton DG, Zderic TW. Role of low energy expenditure and sitting in obesity, metabolic syndrome, type 2 diabetes, and cardiovascular disease. Diabetes. 2007 Nov;56(11):2655-67. doi: 10.2337/db07-0882. Epub 2007 Sep 7. PMID 17827399
- [Background] Chau JY, van der Ploeg HP, Dunn S, Kurko J, Bauman AE. A tool for measuring workers' sitting time by domain: the Workforce Sitting Questionnaire. Br J Sports Med. 2011 Dec;45(15):1216-22. doi: 10.1136/bjsports-2011-090214. Epub 2011 Sep 22. PMID 21947817
- [Background] Cook AJ, Degood DE. The cognitive risk profile for pain: development of a self-report inventory for identifying beliefs and attitudes that interfere with pain management. Clin J Pain. 2006 May;22(4):332-45. doi: 10.1097/01.ajp.0000209801.78043.91. PMID 16691085
- [Background] Waddell G, Newton M, Henderson I, Somerville D, Main CJ. A Fear-Avoidance Beliefs Questionnaire (FABQ) and the role of fear-avoidance beliefs in chronic low back pain and disability. Pain. 1993 Feb;52(2):157-168. doi: 10.1016/0304-3959(93)90127-B. PMID 8455963